CLINICAL TRIAL: NCT00004041
Title: Phase I Trial of Adenovirus-Mediated Wild-Type P53 Gene Therapy for Malignant Gliomas
Brief Title: Gene Therapy in Treating Patients With Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9703; CDR0000066871 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2004-07-19 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — advexin

INTERVENTIONS:
Biological: Ad5CMV-p53 gene
Procedure: conventional surgery

SUMMARY:
RATIONALE: Inserting the gene for adenovirus p53 into a person's tumor may improve the body's ability to fight cancer.

PURPOSE: Phase I trial to study the effectiveness of gene therapy in treating patients who have recurrent malignant gliomas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the biological effects at the molecular level of intratumoral administration of adenovirus p53 gene (Ad-p53) in patients with malignant primary glioma. II. Determine the maximum tolerated dose of intratumoral Ad-p53 in these patients. III. Evaluate the qualitative and quantitative toxicity of intratumoral Ad-p53 in this patient population.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive an initial intratumoral stereotactic injection of adenovirus p53 (Ad-p53) over 10 minutes on day 1. In the absence of unacceptable toxicity resulting from this initial injection, patients then undergo tumor resection and receive a series of 1-minute injections of Ad-p53 into the resected tumor cavity wall on day 4. Cohorts of 3-6 patients receive escalating doses of Ad-p53. If 2 of 3 or 3 of 6 patients experience dose limiting toxicity (DLT) at a particular dose level, escalation ceases and the maximum tolerated dose is defined as the previous dose level. Patients are followed closely for 12 weeks, then every 2 weeks for 8 weeks, then every 4 weeks for 8 weeks, and then every 8 weeks until death.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignant primary glioma Glioblastoma multiforme Anaplastic oligodendroglioma Gliosarcoma Mixed malignant glioma Anaplastic astrocytoma Clear evidence of tumor recurrence or progression by CT or MRI within 2 weeks prior to study after failing prior best surgical resection and radiation Surgically accessible tumor for which resection is indicated Tumors greater than 2.0 cm in diameter Tumor not extending into the ventricular system

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 No evidence of bleeding diatheses Hepatic: SGPT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Bilirubin less than 1.5 mg/dL Renal: BUN less than 1.5 times ULN OR Creatinine less than 1.5 times ULN Cardiovascular: Not specified Pulmonary: Not specified Other: No active uncontrolled infection Must be afebrile (less than 38.0 degrees Celsius) No other unstable or serious medical conditions HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy allowed (at least 2 weeks since prior vincristine, 3 weeks since prior procarbazine, and 6 weeks since prior nitrosoureas) and recovered Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: No prior or concurrent anticoagulants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02-25 (Actual); Primary Completion 2002-07-22 (Actual); Study Completion 2003-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F. Lang, MD, Study Chair — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin